CLINICAL TRIAL: NCT02223104
Title: Randomized Controlled Multicenter Study to Evaluate the Performance of Flexima® Active vs. Sensura® in Patients With Colostomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: BBraun Medical SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OPM-G-H-1301
Record Dates: First submitted 2013-10-25; First posted 2014-08-22 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Colostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sensura (Active Comparator): Ostomy pouch
  Interventions: Device: Flexima Active
- Flexima Active (Experimental): Ostomy pouch
  Interventions: Device: Sensura

INTERVENTIONS:
Device: Flexima Active
  Arms: Sensura
Device: Sensura
  Arms: Flexima Active

SUMMARY:
The purpose of this study is to demonstrate that the performance of Flexima Active is non-inferior to the performance of Sensura.

ELIGIBILITY:
Inclusion Criteria:

* patient is at least 18 years old
* patient having a colostomy with a diameter less than 50 mm for users of midi pouches or having a colostomy with a diameter less than 65 mm for users of maxi pouches
* patient having a colostomy for at least 1 month
* patient using currently a one-piece flat ostomy appliance with closed or drainable bags
* patient using minimum 1 product per day with closed pouches or minimum 1 product every two days with drainable pouches
* patient capable to apply and remove the pouch himself or with the help of a caregiver (except health care professional)
* patient having a mental capacity to participate to the study (i.e. to understand the study and to answer to the questions)
* patient agrees to test Flexima® Active (size midi or maxi, beige) during 14 days and Sensura® (size midi or maxi, beige) during 14 days
* patient covered by social security

Exclusion Criteria:

* patient receiving or having received, within the last month, chemotherapy or radiotherapy
* patient currently suffering from peristomal skin complications (bleeding or red and broken skin at the time of inclusion)
* patient currently receiving or having received within the past three weeks systemic or local steroid medication in the peristomal skin
* patient already participating in another clinical study or who have previously participated in this investigation
* pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Level of leakage under the skin protector of Flexima Active in comparison with level of leakage under the skin protector of Sensura. | Up to one day for closed pouches and up to two days for drainable pouches.
  The patient will evaluate the level of leakage under the skin protector after each removal of pouch.
  A 4 scale level will be used:
  * "no leakage under the skin protector",
  * "leakage under the skin protector not soiling clothes",
  * "leakage under the skin protector soiling clothes",
  * "sudden and massive leakage under the skin protector".

SECONDARY OUTCOMES:
Assessment of the condition of peristomal skin | At V1 and V2 protocol visits (at day 0 and day 14)
Acceptability of each pouch | At each protocol visit (day 0, day 14 and day 28)
  Acceptability is defined by those criteria:
  Wearing comfort, Flexibility, Conformability (skin protector adaptation to the skin relief), Ease of handling (pouch application and pouch removal), Tack (immediate adhesivity to the skin after application), Adhesivity (during wear time), Residues on the skin after pouch removal, Filter performance (odours neutralization, limitation of ballooning of the bag), Security feeling with skin protector, Overall security feeling, Overall satisfaction with skin protector, Overall satisfaction with the appliance
Preference between Flexima® Active and Sensura® | At each protocol visits (at day 0, day 14 and day 28)
Assessment of the quality of life with Stoma-QoL questionnaire | At each protocol visits (at day 0, day 14 and day 28)
Adverse(s) Event(s) | At each protocol visits (at day 0, day 14 and day 28)

CONTACTS AND LOCATIONS:
Locations (1):
- Bichat Hospital, Paris, France